CLINICAL TRIAL: NCT04739410
Title: Effectiveness of Ivermectin in SARS-CoV-2/COVID-19 Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: FMH College of Medicine and Dentistry (Other)
Responsible Party: Principal Investigator, Aijaz Zeeshan Khan Chachar, Consultant Physician (Senior Registrar), FMH College of Medicine and Dentistry
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB#FMH-07-2020-IRB-766-M
Record Dates: First submitted 2021-02-02; First posted 2021-02-04 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Covid19
Keywords: Corona virus; SARS-COv-2; Ivermectin; pandemic; antiviral
MeSH Terms: conditions — COVID-19 | interventions — Ivermectin

STUDY DESIGN:
Intervention Model Description: Response of the patients after Ivermectin prescription and response of the patients without Ivermectin prescription was recorded. Response was recorded on the basis of clinical parameters (Fever, Cough, sore throat, Headache, Shortness of breath, lethargy, and fatigue. Any side effects noted after prescription of Ivermectin was recorded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Ivermectin (Experimental): Ivermectin Prescribing protocol: Participants were prescribed Ivermectin 12mg stat per oral and then 12 mg per oral after 12 hours and 12mg per oral after 24 hours and we looked at the response at day 7 on follow up in terms of improvement of symptoms like (Fever, Cough, sore throat, Headache, Shortness of breath, lethargy, and fatigue. and any side effects of the drugs were noted as well.
  Interventions: Drug: Ivermectin
- SOC standard of care (Placebo Comparator): These participants were given standard of care without Ivermectin standard of care only symptomatic treatment
  Interventions: Drug: Ivermectin

INTERVENTIONS:
Drug: Ivermectin — Ivermectin Prescribing protocol: Participants were prescribed Ivermectin 12 mg per oral stat and then 12 mg per oral after 12 hours and 12 mg per oral after 24 hours and we looked at the response at day 7 on follow up in terms of improvement of symptoms like (Fever, Cough, sore throat, Headache, Shortness of breath, lethargy, and fatigue.Any side effects of the drugs were noted as well
  Other Names: Experimental

SUMMARY:
Background:

The first case of Infection with severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) were diagnosed in Wuhan, China in 2019. In the first half of 2020 this disease has already converted into a global pandemic. Objectives: To assess the efficacy of Ivermectin in mild cases of COVID-19 patients on the basis of predefined assessment criteria. Study Settings: Fatima Memorial Hospital, Lahore Study Design: Open label randomized control trial. Duration of Study: From 1st May, 2020 to 30th June, 2020.Patients & Methods: Sample size and technique: Sample size was 50 patients; 25 patients were kept in control group and 25 patients were kept in experimental group

DETAILED DESCRIPTION:
The first case of Infection with severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) were diagnosed in Wuhan, China in 2019. In the first half of 2020 this disease has already converted into a global pandemic, having different forms of presentation in different patients.

Exponential rise in its cases along with associated mortality has shaken the world.

The severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) is a single-stranded ribonucleic acid (RNA) virus that causes a severe acute respiratory syndrome. The virus was originally called SARS-CoV-2 named officially by World Health Organization as COVID-19 and a global health emergency. The first known case of infection was recorded in early December 2019 and subsequently spread to various continents, including Europe and the United States.Generally, 75 percent of patients recover without any notable complication however 25 percent can experience associated complications leading to intensive care unit transfer and even mortality.

Ivermectin has different effects to treat variety of diseases and it has proven antimicrobial, antiviral, and anti-cancer properties and considered as a wonder drug. It is highly effective against many microorganisms including some viruses. Many studies revealed its antiviral effects on RNA viruses such as Zika, dengue, yellow fever, West Nile, Hendra, Newcastle, Venezuelan equine encephalitis, chikungunya, Semliki Forest, Sindbis, Avian influenza A, Porcine Reproductive and Respiratory Syndrome, Human immunodeficiency virus(HIV) type 1, and severe acute respiratory syndrome coronavirus SARS-CoV-2. Fon other hand there are few studies showing antiviral effects of ivermectin against DNA viruses such as Equine herpes type 1, BK polyomavirus, pseudorabies, porcine circovirus 2, and bovine herpesvirus 1.5 Ivermectin plays a vital role in several biological mechanisms, therefore it could emerge as a potential candidate in the treatment of a wide range of viruses including COVID-19 as well as other types of positive-sense single-stranded RNA viruses. In vivo studies of animal models revealed a broad range of antiviral effects of ivermectin, however, more clinical trials are necessary as it's the need of the hour to do so, as we can validate the potential efficacy of ivermectin in clinical settings.

The recent report by Caly et al.6 describing the antiviral potential of ivermectin against the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) in vitro arrive to the agenda of potential candidates for COVID-19 treatment.

Currently, there is not any Food and drug administration (FDA) approved specific effective antiviral treatment available for COVID-19.Although most of the COVID-19 patients have mild or moderate courses, up to 5%-10% can have severe, potentially life threatening course, there is an urgent need for development of effective & safe drugs to deal with this novel virus. Optimized supportive care remains the mainstay of therapy. There are more than 300 clinical trials going on, various antiviral and immunomodulating agents are in different stages of evaluation for COVID-19 in those trials and results/ primary end points of few trials will be published in the next couple of months. Despite the urgent need to find an effective and safe antiviral treatment for COVID-19 through randomized controlled studies, certain agents are being used all over the world based on either in-vitro or conclusive evidence or observational studies.

The clinical efficacy and utility of ivermectin in SARS-CoV-2-infected patients is unpredictable at this stage, as we are dealing with a completely novel virus.

There is an urgent need for investigation of the mortality causes and development of novel therapeutic options for severe COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* All patients diagnosed with COVID-19 infection with positive reverse transcriptase RT-PCR test, who were willing to participate in this study
* Patients having age of 18-75 years
* Patients of both genders male and female
* Patients who had mild symptoms of Corona virus disease and RT- PCR positive for SARS-Cov-2
* Ability to take oral medication and were willing to adhere to the drug intake regimen

Exclusion Criteria:

* Known severe allergic reactions to Ivermectin
* Pregnancy or breastfeeding
* Severe symptoms likely attributed to Cytokine Release Storm
* Malignant diseases
* Chronic kidney disease
* Cirrhosis liver with Child class B or C

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Resolution of symptoms | 7 days
  Will look for resolution of Fever, Fatigue, myalgias, cough and we had an questionaire for that as well and followed up on their chest x rays for progression of the disease
Progression of the disease | 14 days
  did the disease progress from mild to moderate severity, like follow up chest x ray showed more infiltrates or their oxygen saturations in % dropped from their baseline and baseline symptoms persisted and got worse

CONTACTS AND LOCATIONS:
Overall Officials: Aijaz Zeeshan Khan Chachar, MBBS,FCPS, Principal Investigator — FMH College of Medicine & Dentistry
Locations (1):
- Aijaz Zeeshan Khan Chachar, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
whatever is needed, will share if needed at any time
Supporting Information: Study Protocol, SAP, ICF
Time Frame: as soon as i will have time to respond